CLINICAL TRIAL: NCT05841381
Title: Adjuvant Study of Pyrotinib in Combination With Trastuzumab in Patients With HER2 Positive and Lymph Node Negative Invasive Breast Cancer
Brief Title: Adjuvant Study of Pyrotinib in Combination With Trastuzumab in HER2 Positive Invasive Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC
Record Dates: First submitted 2023-04-22; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- arm 1 (Experimental): Pyrotinib Plus trastuzumab and paclitaxel
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Paclitaxel
- arm 2 (Active Comparator): trastuzumab and paclitaxel
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pyrotinib — pyrotinib: 400mg orally daily for 1 year
  Arms: arm 1
Drug: Trastuzumab — 8mg/kg iv load followed by 6mg/kg iv 3-weekly for a total of 17 cycles
Drug: Paclitaxel — 80mg/m2 per week for a total of 12 weeks

SUMMARY:
This is an open label, phase III study evaluating the efficacy and safety of Pyrotinib in Combination With Trastuzumab and paclitaxel in patients HER2 Positive and lymph node negative invasive Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Females 18-70 years old;
* Pathological confirmed of stage I-II breast cancer: histologically confirmed that the longest diameter of invasive cancer is no less than 1cm and no more than 5cm and the lymph node is negative (N0);
* The pathological type of immunohistochemistry must meet the following conditions: HER-2 (3+) or HER-2 (0-2 +) with FISH detection is amplified;
* For patients with invasive lesions on both sides, if both lesions are HER-2 positive and meet the tumor size requirements, then can be enrolled;
* Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN#and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula);
* LVEF>50%;
* The patient voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

* Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy;
* Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ;
* Has metastic (Stage 4) breast cancer;
* Pregnant or breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
* Patients participating in other clinical trials at the same time;
* Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmHg, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
* Has severe or uncontrolled infection;
* Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders;
* The researchers considered patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2023-05-06 (Estimated); Primary Completion 2028-05-06 (Estimated); Study Completion 2033-05-06 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 year

SECONDARY OUTCOMES:
distant recurrence free survival | 5 year
overall survival | 5 year
adverse effects | 5 year

IPD SHARING:
Plan to Share IPD: No